CLINICAL TRIAL: NCT00539110
Title: Differential Effects of Zolpidem Versus Ramelteon on Nocturnal Sleep in Pediatric Burn Patients: A Prospective, Randomized Crossover Trial With Polysomnographic Recordings
Brief Title: Differential Effects of Zolpidem Versus Ramelteon in Burned Children
Acronym: Sleep3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Director, Nutrition Services, Shriners Hospitals for Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-04-07-01
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Sleep; Burns
MeSH Terms: conditions — Burns | interventions — Zolpidem; ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zolpidem (Experimental): zolpidem or ramelteon dosed at 2200 and 0200 per feeding tube depending on randomization
  Interventions: Drug: zolipidem
- ramelteon (Active Comparator): ramelteon or zolpidem dosed at 2200 and 0200 per the feeding tube depending on randomization
  Interventions: Drug: ramelteon

INTERVENTIONS:
Drug: zolipidem — zolpidem dosed at 2200 and 0200 per feeding tube depending on randomization
  Other Names: Ambien
  Arms: zolpidem
Drug: ramelteon — ramelteon dosed at 2200 and 0200 per feeding tube depending on randomization
  Other Names: rozerem
  Arms: ramelteon

SUMMARY:
To examine sleep changes following therapeutic drug interventions designed to promote sleep.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury > 20% total body surface area
* Between 3 and 18 years of age
* < 7 days from acute injury
* Written informed consent and HIPPA release signed

Exclusion Criteria:

* Suspected anoxic brain injury or head injury
* Hepatic or endocrine disease
* History of alcoholism or substance abuse
* Pre-existing neurological or primary psychiatric disorder
* Medical history of pre-existing sleep disorder or lactose deficiency
* Questionable survival (<72 hrs) as decided by PI
* Receipt of drugs with known effects on sleep within 24 hrs of study entry
* No informed consent/HIPPA release

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gottschlich, PhD, Principal Investigator — Shriners Hospital for Children
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stockmann C, Spigarelli MG, Healy DP, Gottschlich MM, Kagan R, Balch AH, Sherwin C. Application of a method used to deconstruct a single dose pharmacokinetic profile from multiple dose data. Biopharm Drug Dispos. 2015 Sep;36(6):405-409. doi: 10.1002/bdd.1949. Epub 2015 Apr 21. PMID 25766031
- [Background] Stockmann C, Gottschlich MM, Healy D, Khoury JC, Mayes T, Sherwin CM, Spigarelli MG, Kagan RJ. Relationship between zolpidem concentrations and sleep parameters in pediatric burn patients. J Burn Care Res. 2015 Jan-Feb;36(1):137-44. doi: 10.1097/BCR.0000000000000164. PMID 25185933
- [Background] Stockmann C, Sherwin CM, Buterbaugh W, Spigarelli MG, Gottschlich MM, Healy D, Kagan RJ. Preliminary assessment of zolpidem pharmacokinetics in pediatric burn patients. Ther Drug Monit. 2014 Jun;36(3):295-301. doi: 10.1097/FTD.0000000000000017. PMID 24365985

RESULTS

PARTICIPANT FLOW:
Groups:
- Zolpidem First, Then Ramelteon: medication dosed at 2200 and 0200 per feeding tube
  washout with no sleep meds (3 nights); zolpidem (x4 nights); washout (x3 nights); then ramelteon (x4 nights)
- Ramelteon, Then Zolpidem: medication dosed at 2200 and 0200 per the feeding tube
  washout with no sleep meds (x3 nights); ramelteon (x4 nights); washout (x3 nights); then zolpidem (x 4 nights)
Period: Overall Study
Arm/Group | Zolpidem First, Then Ramelteon | Ramelteon, Then Zolpidem
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were ten patients total, crossover design, so each of the 10 patients received both zolpidem and ramelteon.
  Mean age 7.8 years
Groups:
- Zolpidem First, Then Ramelteon; Ramelteon First, Then Zolpidem: dosed at 2200 and 0200 per the feeding tube
- Total: Total of all reporting groups
Arm/Group | Zolpidem First, Then Ramelteon | Ramelteon First, Then Zolpidem | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (1.6) | 7.8 (1.6) | 7.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Polysomnography Data
Description: Determine if intervention product elicits more total sleep time
Time Frame: 2 weeks postburn
Measure: Mean (Standard Error); unit: minutes
Groups:
- Zolpidem: medication dosed at 2200 and 0200 per feeding tube
- Ramelteon: dosed at 2200 and 0200 per the feeding tube
Arm/Group | Zolpidem | Ramelteon
Number analyzed (Participants) | 6 | 6
minutes | 373 (40) | 346 (33)

2. Secondary Outcome: Pharmacokinetics
Description: evaluate the PK of zolpidem following standard dosing practices
Time Frame: 2 weeks postburn
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Zolpidem: medication dosed at 2200 and 0200 per feeding tube
  zolipidem: dosed at 2200 and 0200 per feeding tube
- Ramelteon: dosed at 2200 and 0200 per the feeding tube
  ramelteon: medication dosed at 2200 and 0200 per feeding tube
Arm/Group | Zolpidem | Ramelteon
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes